CLINICAL TRIAL: NCT02338102
Title: Nasal Saline Irrigation After Radiation Therapy for Oropharyngeal Cancer: A Pilot Study
Brief Title: Nasal Saline Irrigation After Radiation Therapy for Oropharyngeal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Shnayder (Other)
Responsible Party: Sponsor-Investigator, Lisa Shnayder, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000087
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Nasal Obstruction; Rhinitis, Vasomotor; Epistaxis
MeSH Terms: conditions — Nasal Obstruction; Rhinitis, Vasomotor; Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Subjects in this group will perform twice daily nasal irrigations. Nasal irrigations will be performed by using premeasured salt packets mixed with distilled water in NeilMed irrigation bottles. The subject will be instructed to lean forward over the sink, place the bottle up to the nostril, and hold their breath while gently squeezing the bottle. One bottle is used to irrigate both nostrils, using half the solution on each side.
  Interventions: Other: Saline mixture
- Control Group (No Intervention): Subjects randomized to this arm receive no intervention.

INTERVENTIONS:
Other: Saline mixture — premeasured salt packets mixed with distilled water
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to learn whether nasal saline irrigation is beneficial to patients undergoing radiation therapy for oropharyngeal cancer.

DETAILED DESCRIPTION:
In this study, subjects are randomized to one of two study arms. They are either randomized to receive nasal saline irrigation treatment (treatment group) or not to receive any nasal irrigation treatment (control group). Subjects randomized to the treatment group will be provided with saline packets to mix with water. All study subjects will be asked to complete questionnaires during the study. If a subject completes all study related activities, their total length of participation in the study will last about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the KUMC Ear, Nose and Throat clinic with oropharyngeal cancer that have undergone radiation therapy as the primary treatment

Exclusion Criteria:

* Patients that are at high risk for infection secondary to nasal irrigation
* Patients with autoimmune disease or immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in quality of life, measured using Sino-Nasal Outcome Test (SNOT-20) summary scores | Change from Baseline to Month 2
  Outcome measured using Sino-Nasal Outcome Test (SNOT-20) summary scores. Scores will be collected at the baseline visit and again on the Month 2 visit. Outcome represented as a change in mean summary scores between the two visits. Scores can range from 0-5 with 0 being the best and 5 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Yelizaveta Shnayder, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States